CLINICAL TRIAL: NCT00633464
Title: Randomized Phase II Study of Ixabepilone Alone and Ixabepilone Plus Cetuximab as First-Line Treatment for Female Subjects With Triple Negative (ER, PR, Her2 Negative) Locally Advanced Non-resectable and/or Metastatic Breast Cancer
Brief Title: Randomized Phase II Study of Ixabepilone Alone and Ixabepilone Plus Cetuximab as First-Line Treatment for Female Subjects With Triple Negative Locally Advanced Non-resectable and/or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-139
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Results first posted 2012-04-24 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Triple Negative Locally Advanced Non-resectable Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (ixabepilone 40 mg^2) (Experimental): ixabepilone 40 mg/m^2 every 3 weeks
  Interventions: Drug: ixabepilone
- Arm B (cetuximab 250 mg/m^2 + ixabepilone 40 mg/m^2) (Experimental): cetuximab 400 mg/m^2 loading dose then 250 mg/m^2 weekly + ixabepilone 40 mg/m^2 every 3 weeks
  Interventions: Drug: ixabepilone + cetuximab

INTERVENTIONS:
Drug: ixabepilone — injection, intravenous (IV), until unacceptable toxicity or progression or 15 months after the Last Subject First Visit (LSFV), whichever comes first.
  Ixabepilone 40 mg/m^2 was administered as a 3-hour IV continuous infusion on Day 1 in a 21-day cycle provided the participant met the re-treatment criteria.
  Other Names: IXEMPRA; BMS-247550
  Arms: Arm A (ixabepilone 40 mg^2)
Drug: ixabepilone + cetuximab — Ixabepilone: injection, IV, until unacceptable toxicity or progression or 15 months after the LSFV, whichever comes first.
  Ixabepilone 40 mg/m^2 was administered as a 3-hour IV continuous infusion on Day 1 in a 21-day cycle provided the participant meets the re-treatment criteria.
  Cetuximab: injection, IV, until unacceptable toxicity or progression or 15 months after the LSFV, whichever comes first.
  Cetuximab 400 mg/m^2 was administered as a 2-hour IV loading dose via in-line filtration with an infusion pump, gravity drip, or a syringe pump on Day 1 of first cycle then 250 mg/m^2 1-hour IV once a week, i.e. on Days 1, 8, and 15 of each cycle provided the participant meets the re-treatment criteria.
  Other Names: IXEMPRA; BMS-247550; ERBITUX; BMS-564717
  Arms: Arm B (cetuximab 250 mg/m^2 + ixabepilone 40 mg/m^2)

SUMMARY:
The purpose of this study was to estimate the response rate of ixabepilone monotherapy, and the combination of ixabepilone plus cetuximab as first-line treatment of female subjects with triple negative (estrogen receptor [ER], progesterone receptor [PR], Human Epidermal Growth Factor Receptor 2 [HER2] negative) locally advanced non-resectable and/or metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with triple negative (ER, PR, and HER2 negative) locally advanced non-resectable and/or metastatic breast cancer
* Prior adjuvant or neoadjuvant anthracycline-based chemotherapy

Exclusion Criteria:

* Tumors that are fluorescence in situ hybridization test (FISH) positive or immunohistochemistry (IHC) 3+
* Neuropathy > Grade 1
* Prior systemic therapy for metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- Austria (2):
  - Local Institution, Graz
  - Local Institution, Vienna
- Czechia (2):
  - Local Institution, Brno
  - Local Institution, Prague
- France (7):
  - Local Institution, Bayonne
  - Local Institution, Dijon
  - Local Institution, Lyon
  - Local Institution, Paris
  - Local Institution, Saint-Brieuc
  - Local Institution, Saint-Herblain
  - Local Institution, Toulouse
- Local Institution, Thessaloniki, Greece
- Local Institution, Napoli, Italy
- Poland (2):
  - Local Institution, Gdansk
  - Local Institution, Olsztyn
- Local Institution, Barcelona, Spain

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixabepilone 40 mg/m^2: ixabepilone 40 mg/m^2 every 3 weeks
- Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2: cetuximab 400 mg/m^2 loading dose then 250 mg/m^2 weekly + ixabepilone 40 mg/m^2 every 3 weeks
Period: Overall Study
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2
Started | 40 | 39
Treated | 40 | 37
Completed | 40 (Completed=Offstudy;major reasons:Disease progression-27,study drug toxicity-7,max clinical benefit-3) | 37 (Completed=Offstudy;major reasons:Disease progression-25,study drug toxicity-4,subject request-3)
Not Completed | 0 | 2
Not completed — Never Treated (Not met study criteria) | 0 | 1
Not completed — Never Treated (Randomized in error) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2 | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Customized [Median (Full Range); unit: years] | 53.0 [29.0 to 75.0] | 50.0 [31.0 to 79.0] | 53.0 [29.0 to 79.0]
Age, Customized [Number; unit: participants]
  < 65 | 35 | 32 | 67
  >=65 | 5 | 7 | 12
Sex/Gender, Customized [Number; unit: participants]
  Female | 40 | 39 | 79
Race/Ethnicity, Customized [Number; unit: participants]
  White | 39 | 39 | 78
  Black/African American | 1 | 0 | 1
Karnofsky Performance Status [Number; unit: participants] — Karnofsky Performance Status classifies patients according to their functional impairment. Scores range from 0-100 units on a scale, the lower the score, the worse the survival for most serious illnesses.
  100: Normal, no complaints; 90: Able to carry on normal activities; minor signs or symptoms of disease; 80: Normal activity with effort; some signs or symptoms of disease.
  participants
    100 | 23 | 23 | 46
    90 | 6 | 5 | 11
    80 | 11 | 10 | 21
    Not Reported | 0 | 1 | 1
Setting of Prior Chemotherapy [Number; unit: participants] — Participants may have received chemotherapy in more than one setting.
  participants
    Adjuvant therapy | 28 | 22 | 50
    Neo-adjuvant therapy | 20 | 20 | 40
    Adjuvant and Neo-adjuvant | 8 | 3 | 11

OUTCOME MEASURES:

1. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time interval from date of randomization until the first date of documented progressive disease (PD) or death from any cause without prior documentation of progression. The PFS was estimated using the Kaplan-Meier product-limit method, and a two-sided 95% CI for the median PFS time was computed using the method of Brookmeyer and Crowley.
  PD: At least 20% increase in sum of LD of target lesions in reference to smallest sum LD recorded at or following baseline or unequivocal progression of existing non-target lesion(s) overall.
Time Frame: From the date of randomization to date of progression, death, or last tumor assessment (maximum participant PFS of 17 months)
Population: All randomized participants. Participants who did not progress or die were censored on the date of their last tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 40 | 39
months | 4.1 [3.0 to 4.9] | 4.1 [2.7 to 6.1]

2. Secondary Outcome: Time to Response
Description: Time to response is defined as the time from the date of start of treatment until measurement criteria are first met for PR or CR (whichever is recorded first).
  CR: Disappearance of all target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the LD of all target lesions with reference to the baseline sum LD.
  Time to response was estimated using the Kaplan-Meier product-limit method.
Time Frame: Assessed every 6 weeks for first 12 months from randomization thereafter every 3 months until CR or PR (maximum participant time to response of 18.3 weeks.)
Population: Randomized participants with response of CR or PR.
Measure: Median (Full Range); unit: weeks
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 12 | 14
weeks | 8.8 [5.1 to 12.0] | 6.5 [5.1 to 18.3]

3. Primary Outcome: Percentage of Participants With Objective Response (OR; Using Response Evaluation Criteria in Solid Tumors [RECIST])
Description: The participant had an OR if her best overall response (BOR) during the study was either a complete response (CR) or a partial response (PR) according to the RECIST as determined by the investigator. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (LD) of all target lesions. Confidence interval (CI) was Computed using Clopper-Pearson method.
Time Frame: Assessed every 6 weeks for first 12 months from randomization thereafter every 3 months until disease progression (maximum participant objective response of 18.3 weeks)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 40 | 39
percentage of participants | 30.0 [16.6 to 46.5] | 35.9 [21.2 to 52.8]

4. Secondary Outcome: Duration of Response
Description: Defined as period from the time that measurement criteria are first met for CR or PR until first date of documented PD or death. Estimated using the Kaplan-Meier product-limit method; CI was computed using Brookmeyer and Crowley method. CR: Disappearance of all target and non-target lesions. PR: At least 30% reduction from baseline in the sum of LD of all target lesions with reference to baseline sum LD. PD: At least 20% increase in sum of LD of target lesions in reference to smallest sum LD recorded at or following baseline or unequivocal progression of existing non-target lesion(s) overall.
Time Frame: From the date of first PR or CR assessment to date of progression, death, or last tumor assessment (maximum participant duration of response of 15.6 months)
Population: Randomized participants with response of CR or PR. Participants who did not relapse or die were censored on the date of their last tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 12 | 14
months | 4.5 [3.0 to 8.7] | 4.5 [3.4 to 6.9]

5. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Adverse Events (AEs), and AEs Leading to Discontinuation of Study Therapy Per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0
Description: AE: New untoward medical occurrence or worsening of a preexisting medical condition that does not have causal relationship with this treatment. SAE: Untoward medical event that at any dose: results in death, persistent or significant disability/incapacity, drug dependency/abuse; life-threatening, an important medical event, a congenital anomaly/birth defect; requires inpatient hospitalization/prolongs existing hospitalization. Grade (GR) 3=Severe; and GR4=Life-threatening or disabling. Other reasons for death included hepatic failure and respiratory distress.
Time Frame: Assessed from the date of first dose until at least 30 days after the last dose of study drug. Median time on ixapebilone therapy was 15 weeks (range: 3-54 weeks for ixabepilone arm; 3-36 weeks for ixabepilone+cetuximab arm)
Population: All treated participants: Participants who received any treatment (ixabepilone or cetuximab).
Measure: Number; unit: participants
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 40 | 37
participants
  All Deaths | 8 | 9
  Deaths due to Disease Progression | 8 | 7
  Deaths due to Other Reasons | 0 | 2
  At least one SAE (Any Grade) | 9 | 12
  At least one SAE (Grade 3 to 4) | 4 | 11
  At least one Related SAE (Any Grade) | 3 | 6
  At least one Related SAE (Grade 3 to 4) | 2 | 6
  At least one AE (Any Grade) | 40 | 37
  At least one AE (Grade 3 to 4) | 21 | 25
  At least one Related AE | 37 | 37
  At least one Related AE (Grade 3 to 4) | 18 | 22
  AEs leading to discontinuation (Any Grade) | 8 | 13
  AEs leading to discontinuation (Grade 3 to 4) | 3 | 7

6. Secondary Outcome: Number of Participants With Hematology Abnormalities
Description: Grading: NCI CTCAE, Version 3.0. GR1=mild, GR2=moderate, GR3=severe, GR4=life threatening or disabling. Normal ranges provided by local laboratory and may also vary by age and sex. Hemoglobin:GR1=<LLN-10.0g/dL; GR2=<10.0-8.0g/dL; GR3:<8.0-6.5g/dL, GR4:<6.5g/dL. Platelets:GR1=<LLN-75.0*10^9/L; GR2=<75.0-50.0*10^9/L; GR3:<50.0-25.0*10^9/L, GR4:<25.0*10^9/L. Absolute Neutrophil Count (ANC):GR1=<LLN-1.5*10^9 /L; GR2=<1.5-1.0*10^9/L; GR3:<1.0-0.5*10^9/L; GR4:<0.5*10^9/L. White blood cell (WBC):GR1=<LLN-3.0*10^9/L; GR2=<3.0-2.0*10^9/L; GR3:<2.0-1.0*10^9/L; GR4:<1.0*10^9/L. LLN=lower limit of normal.
Time Frame: Assessed prior to 1st cycle, at beginning of each cycle, weekly (cetuximab treatment), and every 4 weeks within 30 days after last dose of study drug. Median time on ixapebilone therapy: 15 weeks (range:3-54:ixabepilone arm;3-36:ixapebilone+cetuximab arm)
Population: Treated participants: Participants who received any treatment (ixabepilone or cetuximab). n=number of participants with measures available at the time.
Measure: Number; unit: participants
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 40 | 37
participants
  White Blood cell (WBC) GR 1-4 | 33 | 34
  WBC GR 3-4 | 13 | 16
  Absolute Neutrophil Count(ANC) GR 1-4 (n=39; n=37) | 33 | 31
  ANC GR 3-4 (n=39; n=37) | 19 | 18
  Platelet Count GR 1-4 (n=39; n=37) | 11 | 4
  Platelet Count GR 3-4 (n=39; n=37) | 0 | 0
  Hemoglobin GR 1-4 | 29 | 27
  Hemoglobin GR 3-4 | 0 | 0

7. Primary Outcome: Number of Participants With Best Overall Response as Assessed With Response Criteria in Solid Tumors (RECIST)
Description: PD = At least a 20% increase in the sum of LD of target lesions in reference to the smallest sum LD recorded at or following baseline or unequivocal progression of existing non-target lesion(s) overall; Stable Disease (SD) = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (LD) of all target lesions.
Time Frame: Assessed at 6 week intervals for first 12 months from randomization, thereafter every 3 months (to a maximum follow-up for tumor response of 17 months).
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 40 | 39
participants
  Complete Response | 3 | 0
  Partial Response | 9 | 14
  Stable Disease | 17 | 12
  Progressive Disease | 9 | 10
  Never Treated | 0 | 2
  Unable to determine | 2 | 1

8. Secondary Outcome: Number of Participants With Serum Chemistry Abnormalities
Description: Grading: NCI CTCAE, Version 3.0. GR1=mild, GR2=moderate, GR3=severe, GR4=life threatening or disabling. Normal ranges provided by local laboratory and may also vary by age and sex. Alanine aminotransferase, aspartate aminotransferase, and alkaline phosphatase: GR1=>ULN-2.5*ULN (upper limit of normal); GR2=>2.5-5.0*ULN; GR3=>5.0-20.0*ULN; GR4:>20.0*ULN. Total bilirubin:GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3-10*ULN, GR4=>10*ULN. Creatinine: GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3.0-6.0*ULN, GR4=>6.0*ULN.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2
Number analyzed (Participants) | 40 | 37
participants
  Alkaline Phosphatase (ALP) GR 1-4 (n=38; n=35) | 9 | 17
  ALP GR 3-4 (n=38; n=35) | 0 | 1
  Alanine Aminotransferase (ALT) GR 1-4 (n=39; n=35) | 10 | 18
  ALT GR 3-4 (n=39; n=35) | 1 | 0
  Aspartate Aminotransferase (AST) GR1-4(n=39; n=35) | 11 | 17
  AST GR 3-4 (n=39; n=35) | 1 | 3
  Total Bilirubin GR 1-4 (n=39; n=35) | 1 | 3
  Total Bilirubin GR 3-4 (n=39; n=35) | 1 | 0
  Creatinine GR 1-4 (n=40; n=36) | 3 | 1
  Creatinine GR 3-4 (n=40; n=36) | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed from the date of first dose until at least 30 days after the last dose of study drug (Median number of ixabepilone cycles were 5 [range: 1-18 cycles for ixabepilone arm; 1-12 cycles for cetuximab + ixabepilone arm])
Arm/Group | Ixabepilone 40 mg/m^2 | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2
Serious Adverse Events (participants affected / at risk) | 9/40 | 12/37
Other Adverse Events (participants affected / at risk) | 40/40 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone 40 mg/m^2 (N=40) | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2 (N=37)
PYREXIA (General disorders) | 2 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
CHEST PAIN (General disorders) | 0 | 1
THROMBOPHLEBITIS (Vascular disorders) | 1 | 0
FATIGUE (General disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ASTHENIA (General disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HAEMORRHAGE (Vascular disorders) | 1 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SKIN INFECTION (Infections and infestations) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INFLAMMATION (General disorders) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 5
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
SINUS ARRHYTHMIA (Cardiac disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone 40 mg/m^2 (N=40) | Cetuximab 250 mg/m^2 + Ixabepilone 40 mg/m^2 (N=37)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 | 8
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 | 4
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 | 10
HEADACHE (Nervous system disorders) | 4 | 9
LACRIMATION INCREASED (Eye disorders) | 2 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 6 | 9
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
PYREXIA (General disorders) | 3 | 12
RASH (Skin and subcutaneous tissue disorders) | 2 | 12
STOMATITIS (Gastrointestinal disorders) | 3 | 3
VOMITING (Gastrointestinal disorders) | 15 | 11
WEIGHT DECREASED (Investigations) | 2 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 8
ACNE (Skin and subcutaneous tissue disorders) | 0 | 15
ALOPECIA (Skin and subcutaneous tissue disorders) | 23 | 13
CHEST PAIN (General disorders) | 4 | 2
CONSTIPATION (Gastrointestinal disorders) | 10 | 12
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 | 15
DYSGEUSIA (Nervous system disorders) | 5 | 7
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 2
MUCOSAL INFLAMMATION (General disorders) | 7 | 8
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
NASOPHARYNGITIS (Infections and infestations) | 2 | 2
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 | 10
DEPRESSION (Psychiatric disorders) | 1 | 3
DYSPEPSIA (Gastrointestinal disorders) | 1 | 4
DYSPHAGIA (Gastrointestinal disorders) | 2 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 3
FATIGUE (General disorders) | 8 | 8
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
NEUROPATHY PERIPHERAL (Nervous system disorders) | 3 | 1
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 | 6
ANXIETY (Psychiatric disorders) | 4 | 5
ASTHENIA (General disorders) | 17 | 20
BREAST PAIN (Reproductive system and breast disorders) | 2 | 1
BRONCHITIS (Infections and infestations) | 2 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 | 12
FLUSHING (Vascular disorders) | 2 | 0
HYPERSENSITIVITY (Immune system disorders) | 2 | 2
HYPERTENSION (Vascular disorders) | 3 | 1
INSOMNIA (Psychiatric disorders) | 4 | 6
PAIN (General disorders) | 2 | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 1 | 4
VERTIGO (Ear and labyrinth disorders) | 1 | 3
DIZZINESS (Nervous system disorders) | 2 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 4
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 4
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OEDEMA PERIPHERAL (General disorders) | 1 | 5
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 6
PARONYCHIA (Infections and infestations) | 1 | 2
TACHYCARDIA (Cardiac disorders) | 0 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 2
ANAEMIA (Blood and lymphatic system disorders) | 8 | 8
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 1 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 10
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 2
HOT FLUSH (Vascular disorders) | 3 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 2
NAUSEA (Gastrointestinal disorders) | 13 | 19
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 3
TINNITUS (Ear and labyrinth disorders) | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 4 | 14
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
NEUROTOXICITY (Nervous system disorders) | 2 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 2
PARAESTHESIA (Nervous system disorders) | 3 | 5
RHINITIS (Infections and infestations) | 3 | 5
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 3
CHILLS (General disorders) | 1 | 2
CONJUNCTIVITIS (Eye disorders) | 0 | 3
DRY MOUTH (Gastrointestinal disorders) | 2 | 2
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 0
HYPOTENSION (Vascular disorders) | 0 | 3
LYMPHOEDEMA (Vascular disorders) | 1 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 15 | 6
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 4 | 6
NEUTROPENIA (Blood and lymphatic system disorders) | 18 | 19
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 17 | 17
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.